CLINICAL TRIAL: NCT05782660
Title: Cash Benefits and Reproductive/Perinatal Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sumit Agarwal, Instructor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022P000093-2
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Maternal Care Patterns; Pregnancy Related; Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants in the treatment group received up to $400 per month.
  Interventions: Other: Cash Benefit
- Control Group (Active Comparator): Participants in the control group did not receive monthly cash benefits.
  Interventions: Other: No Cash Benefit

INTERVENTIONS:
Other: Cash Benefit — Spending from the cards was not restricted to food but could be spent on anything and anywhere Visa was accepted. The debit cards were credited with the first payment on November 18th, 2020 and the second payment on December 18th, 2020. The program continued with monthly credits through August 2021.
  Other Names: Basic Income; Debit Card
  Arms: Treatment Group
Other: No Cash Benefit — No monthly cash benefit.
  Arms: Control Group

SUMMARY:
During the first two years of the COVID-19 pandemic, the City of Chelsea, Massachusetts held a lottery to allocate cash benefits to its residents for ten months. Using data from the Chelsea Eats program, the investigators propose to study the impact of the cash benefit on reproductive and perinatal health.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Chelsea, Massachusetts
* Household income at or below 30% of the U.S. Department of Housing and Urban Development's Area Median Income
* Childbearing age

Exclusion Criteria:

* See inclusion criteria

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3615 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | 20 months
  Pregnancies will be identified using the electronic health record, documented with a positive urine or blood pregnancy test, ultrasound, and/or diagnosis codes over the 10 months of the trial; because pregnancy without delivery is the primary outcome for our main analysis, the investigators will then determine whether each pregnancy did or did not result in a live childbirth delivered vaginally or via Cesarean section, which can occur after the 10 months of the trial

SECONDARY OUTCOMES:
Miscarriage | 20 months
  Miscarriages presenting to the health care setting identified using diagnosis codes and documentation within clinical notes
Abortion | 20 months
  Procedural abortions and prescriptions for medical abortions, focusing specifically on induced abortions
Prenatal vitamin prescriptions prior to pregnancy | 10 months
  New use of prenatal vitamins, including multivitamins, as prescribed or documented in the electronic health record
Contraception | 10 months
  Utilization of long-acting reversible contraceptive methods (intrauterine devices or implants) and prescriptions for hormonal birth control methods (pill, patch, ring)
Number and timing of prenatal visits before delivery | 20 months
  Prenatal visits before delivery and initiation during first trimester
Composite of birth outcomes | 20 months
  Following McConnell et al., this outcome is a composite of at least one of: low birth weight, preterm birth, small for gestational age, or perinatal mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sumit D Agarwal, MD, MPH, Principal Investigator — Brigham and Women's Hospital and Harvard Medical School
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT05782660/Prot_SAP_000.pdf